CLINICAL TRIAL: NCT01364792
Title: A Double Blind Placebo Controlled Study of Valaciclovir in Treatment of Psychosis in Patients With Schizophrenia
Brief Title: To Rescue Cognition With Valaciclovir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Hans C Klein, MD, PhD, psychiatrist, Psychiatrist, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Valaciclovir-1
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Schizophrenia; Psychosis
Keywords: schizophrenia; treatment; inflammation; neuroinflammation; hippocampal
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Inflammation; Neuroinflammatory Diseases | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valaciclovir (Experimental): The patients in the experimental group will be treated with 4 times 2 grams valaciclovir per day for seven days.
  Interventions: Drug: Valaciclovir
- Placebo (Placebo Comparator): Patient receives placebo four times a day for seven days.
  Interventions: Drug: Valaciclovir

INTERVENTIONS:
Drug: Valaciclovir — 4 times 2 grams valaciclovir per day, administrated orally, for seven days.
  Other Names: Zelitrex; Anti-viral drugs

SUMMARY:
This is a one-week, randomized, double blind add-on study of valaciclovir versus placebo in 24 clinical patients with Schizophrenia according to DSM IV, currently experiencing psychosis as is defined by the positive items of the Positive and Negative Syndrome Scale (PANNS) score, being five or higher on one item or four on two items of this scale. Each patient will be randomized to double blind treatment with either valaciclovir or placebo for one week.

The main objective is to find a pre- and post-valaciclovir treatment difference in hippocampal inflammation, as measured with positron emission tomography. The secondary objective is to improve cognition by the supposed anti-inflammatory effect on the hippocampus of valaciclovir. This is measured by pre- and post-treatment performance on the PANSS, the attention and memory test.

Both the treatment team and the patient will remain blinded during the course of the study. Following the active treatment phase, patients will receive treatment as clinically indicated.

DETAILED DESCRIPTION:
Rationale:

Schizophrenia is a chronic and disabling brain disease, with unknown aetiology. Recently, we have shown the presence of an inflammatory process in the hippocampus of schizophrenic patients during psychosis. In addition, we found evidence for the presence of herpes viruses in the temporal lobe of schizophrenic patients during psychosis. Taken together, we hypothesize that the hippocampal inflammation is caused by the presence of herpes viruses, and that this inflammation interferes with the normal involvement of the hippocampus in cognition. Anti-viral treatment, with valaciclovir, that reduces the activity herpes viruses in the hippocampus could reduce the neuroinflammation and thus improve cognition and symptoms in schizophrenia.

Objective:

The main objective is to find a pre- and post-valaciclovir treatment difference in hippocampal inflammation, as measured with positron emission tomography, in schizophrenic patients exposed to a psychotic episode. The secondary objective is to improve cognition by the supposed anti-inflammatory effect on the hippocampus of valaciclovir.

Study design:

The study is double-blind randomized placebo-controlled trial. Study population: For this study, 24 male patients compliant with schizophrenia disorder (DSM-IV codes 295.xx) are included that have a psychosis. The age should be above 18 and patients of all ethnic backgrounds can be included.

Intervention (if applicable):

Of the 24 included patients, 12 patients will receive 8 g (4x2 g per day) of valaciclovir daily for a period of 7 consecutive days and 12 patients will receive 8 g (4x2 g per day) of placebo daily for 7 consecutive days.

Main study parameters/endpoints: The main study parameters are the pre-and post-treatment [11C]-PK11195 binding potential (an inflammatory marker) in the hippocampus, the pre- and post-treatment performance on the PANSS, the attention, memory and IQ test.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Patients will be admitted to a psychiatric hospital, if not already admitted as a part of their regular treatment, and treated with valaciclovir for seven consecutive 24-h periods. Patients have to fill in a questionnaire and have to undergo a part of the Schedules for Clinical Assessment in Neuropsychiatry (SCAN) interview and a MRI scan once, and have to undergo a PANSS interview, attention, memory and IQ tests, and PET scan twice. A total of 345 ml of blood will be taken for the determination of kidney and liver function, herpes virus antibodies, acyclovir levels in blood and for the PET scan data-analysis. Treatment with valaciclovir may cause nausea and headache but the risk of serious side effects is low (<1 out of 10.000). For the PET scan, the arterial catheterization can cause discomfort and the patients are exposed to radioactivity with minor to moderate risk. The patients treated with valaciclovir can have direct benefit form the treatment, because it may reduce symptoms. In general, when this study finds evidence for the involvement of herpes viruses in schizophrenia, this can lead to improved treatment of these patients in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Written informed consent for participation
* Diagnosis: schizophrenia, all subtypes (DSM-IV 295.xx)
* Psychosis, characterised by a total score on the positive scale on the PANSS above 14. In addition, a minimal score of 4 or more on an item of the positive scale.

Exclusion Criteria:

* The use of benzodiazepines. Benzodiazepines have affinity for the peripheral benzodiazepine receptor which is the target receptor for [11C]-PK11195 PET and they can thus interfere with the PET study.
* The use of a nonsteroidal antiinflammatory drug or paracetamol in week before the PET scans and during the treatment of valaciclovir
* The use of anticoagulants or having coagulation disorder
* Use of somatic medication which may affect the immune system (e.g. corticoids, anti-inflammatory drugs, immune suppressive drugs)
* Use of any investigational drug
* Current or recent (<1 year) alcohol or substance abuse
* Disturbed kidney function
* Disturbed liver function
* Current or recent (<4 weeks) infectious or inflammatory disease
* Current systemic disease
* Major metabolic disease (diabetes, hyper- or hypothyroidism, Cushing disease or Addison disease)
* Somatic, organic or neurological disorder
* Participation in a scientific research study (<1 year) involving radiation
* Claustrophobia
* Presence of materials in the body that can be magnetized, like:

  * A pacemaker
  * Metal fragments
  * Shunts
  * Artificial heart valves
  * Vascular clips
  * Fixed hearing aid
  * Tattoos containing metal
  * Hair implants
  * Artificial dentures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To find a pre- and post-valaciclovir treatment difference in hippocampal inflammation | 8-15 days
  The main objective is to find a pre- and post-valaciclovir treatment difference in hippocampal inflammation, as measured with positron emission tomography, in schizophrenic patients exposed to a psychotic episode.

SECONDARY OUTCOMES:
To find pre- and post-treatment [11C]-PK11195 binding potential in other brain areas than the hippocampus. | 8-15 days
  Secondary study parameters are the antibodies against common viruses and the pre- and post-treatment [11C]-PK11195 binding potential in other brain areas than the hippocampus. This is also measured by means of PET and MRI
To find whether the patients hae antibodies against common viruses | 8-15 days
  Secondary study parameters are the antibodies against common viruses, measured in the blood samples.
To find a pre- and post-valaciclovir treatment difference in hippocampal inflammation | 8-15 days
  The secondary objective is to improve cognition by the supposed anti-inflammatory effect on the hippocampus of valaciclovir, this will be measured by means of PANSS, the attention, memory and IQ test.

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Schoevers, MD, Prof., Study Chair — University Medical Centre Grongingen
Locations (1):
- University Medical Center Groningen, University of Groningen, Groningen, Provincie Groningen, Netherlands

REFERENCES:
- [Background] Doorduin J, de Vries EF, Willemsen AT, de Groot JC, Dierckx RA, Klein HC. Neuroinflammation in schizophrenia-related psychosis: a PET study. J Nucl Med. 2009 Nov;50(11):1801-7. doi: 10.2967/jnumed.109.066647. Epub 2009 Oct 16. PMID 19837763
- [Background] Yolken RH, Torrey EF, Lieberman JA, Yang S, Dickerson FB. Serological evidence of exposure to Herpes Simplex Virus type 1 is associated with cognitive deficits in the CATIE schizophrenia sample. Schizophr Res. 2011 May;128(1-3):61-5. doi: 10.1016/j.schres.2011.01.020. Epub 2011 Feb 24. PMID 21353483
- [Background] Dickerson FB, Boronow JJ, Stallings CR, Origoni AE, Yolken RH. Reduction of symptoms by valacyclovir in cytomegalovirus-seropositive individuals with schizophrenia. Am J Psychiatry. 2003 Dec;160(12):2234-6. doi: 10.1176/appi.ajp.160.12.2234. PMID 14638597
- [Background] Dickerson FB, Stallings CR, Boronow JJ, Origoni AE, Sullens A, Yolken RH. Double blind trial of adjunctive valacyclovir in individuals with schizophrenia who are seropositive for cytomegalovirus. Schizophr Res. 2009 Feb;107(2-3):147-9. doi: 10.1016/j.schres.2008.10.007. Epub 2008 Nov 12. PMID 19008077